CLINICAL TRIAL: NCT06127914
Title: A Multiphase Project to Improve Use of Responsive Feeding Among Vulnerable Mother-Infant Dyads
Brief Title: Learning Early Infant Feeding Cues
Acronym: LEIFc
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jessica Bahorski, Assistant Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004685
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Responsive Feeding; Infants; Weight Gain Trajectory
MeSH Terms: conditions — Body-Weight Trajectory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LEIFc Intervention (Experimental): There is only 1 arm of this study. All participants will receive the LEIFc intervention.
  Interventions: Behavioral: Learning Early Infant Feeding Cues

INTERVENTIONS:
Behavioral: Learning Early Infant Feeding Cues — The LEIFc intervention includes individualized responsive feeding education and promotion using the SS-OO-PP-RR (or "super," Setting the Stage, Observation and Opportunities to Embed, Problem Solving and Planning, Reflection and Review coaching approach as a guide. An interventionists interacts with mother-infant dyads during a feeding session at infant ages of 1, 2, 3, 4, and 5 months and coaches the mother on responsive feeding. In particular infant cues of hunger and fullness and tips to assist the mother in making decisions regarding feeding her infant. This will begin with milk based feedings (either breastmilk from breast or bottle, or formula from a bottle), and continue through the transition to solid (complementary) foods.

SUMMARY:
The goal of this clinical trial is to learn more about responsive infant feeding (recognizing baby's signs of hunger and fullness) in mothers and infant enrolled in government-funded maternal-child home visiting programs. The main questions it aims to answer are:

* What are the contributors and barriers to use of responsive infant feeding?
* How can we refine an intervention focused on responsive infant feeding (the Learning Early Infant Feeding Cues intervention) so that mothers will like it and learn skills to help their baby be healthy.
* Will the refined intervention improve use of responsive feeding and be feasible and acceptable to mothers and home visiting programs?

Participants will be asked to:

* Participate in focus groups to talk about their experiences feeding their baby.
* Participate in a study to learn about responsive feeding and how to use it with their baby. This study will start when mothers are in their final month of pregnancy and finish when their baby is 6 months old. Participation will include:

  * Having someone come to the family home during a time when the baby is eating (either from the breast or the bottle). The mother will receive information on the baby's signs from an experienced coach.
  * Agreeing to be video recording during the session when the baby is eating.
  * Completing surveys online.

ELIGIBILITY:
Maternal Inclusion Criteria

* Pregnant mother in the 3rd trimester (28 weeks or beyond)
* Enrolled in a government-funded maternal-child home visiting program
* Maternal age 18 years or older
* English or Spanish speaking
* Anticipated to have custody of infant after birth
* Healthy pregnancy, no complications that are anticipated to result in a preterm birth or extended hospital stay for mother or infant

Maternal Exclusion Criteria

* Gave birth to multiple fetuses
* Age less than 18 years
* Not fluent in English or Spanish
* Expected to not have custody of the infant after birth

Infant inclusion criteria

* Born as a singleton (not a twin, triplet, etc.) to a mother enrolled in a maternal-child home visiting program
* Born full term (37 weeks or beyond)

Infant exclusion criteria

* Congenital anomaly that may interfere with infant feeding or growth after birth (i.e., Down Syndrome, cleft lip/palate)
* Born preterm (born prior to 37 weeks)
* NICU stay beyond 48 hours
* Infant diagnosis of failure to thrive
* Supplemental oxygen
* Enteral feeding device used for feedings

Min Age: 2 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Responsive Feeding | Pre (infant age of 2 weeks) and post (infant age of 6 weeks) intervention.
  Subjective (via survey) and objective (via video) measurement of responsive feeding will be collected. Participants will complete the Infant Feeding Questionnaire to provide a subjective measure of responsive feeding. A feeding session will be video recording then coded for instances of infant cues and maternal response to cues to provide an objective measure of responsive feeding.

SECONDARY OUTCOMES:
Infant growth trajectory | Infant age of 2 weeks to 6 months.
  Infant weight-for-length z-score (WLz) will be calculated from infant weight and length measurements obtained at each study visit. The difference in WLz between infant age of 2 weeks and 6 months will be calculated. Infants will be categorized into 3 growth categories: expected growth (WLz SD change between -0.67 and 0.67, rapid growth > or equal to 0.67, or slow growth < or equal to -0.67.
Age of complementary food introduction | weeks or months since birth
  Current infant feeding practices are collected at each study visit. The infant age (in weeks) at which any foods other than breastmilk or formula were given will be tabulated into a variable.
Duration of any breastfeeding | weeks or months since birth
  Current infant feeding practices are collected at each study visit. Duration of any breastfeeding will be tabulated into a variable.

IPD SHARING:
Plan to Share IPD: Undecided
Aggregated dataset of deidentified participant data will be shared with other research. A data use agreement (DUA) will be required. Video data will not be shared.

REFERENCES:
- [Background] Bahorski J, Romano M, McDougal JM, Kiratzis E, Pocchio K, Paek I. Development of an Individualized Responsive Feeding Intervention-Learning Early Infant Feeding Cues: Protocol for a Nonrandomized Study. JMIR Res Protoc. 2023 Feb 28;12:e44329. doi: 10.2196/44329. PMID 36853761